CLINICAL TRIAL: NCT00063583
Title: Pirfenidone: A Novel Anti-Scarring Therapy for Diabetic Nephropathy
Brief Title: Pirfenidone: A New Drug to Treat Kidney Disease in Patients With Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sharma, Kumar, M.D. (Individual)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Kumar Sharma, UCSD
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DK063017-01 (NIH); R01DK063017 (NIH); NCT00105391 (obsolete NCT alias)
Record Dates: First submitted 2003-06-30; First posted 2003-07-02 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus; Diabetic Nephropathy
Keywords: Kidney disease
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Kidney Diseases | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Pirfenidone
- Pirfenidone 1200 mg/day (Experimental): Pirfenidone will be administered at a dose of 1200 mg/day
  Interventions: Drug: Pirfenidone
- Pirfenidone 2400 mg/day (Experimental): Pirfenidone will be administered at 2400 mg/day
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone will be administered orally at 1200 or 2400 mg day in divided doses

SUMMARY:
The purpose of this study is to determine whether a new investigational drug, pirfenidone, will be an effective therapy for diabetic patients with kidney dysfunction. Our hypothesis is that administration of pirfenidone to type 1 and type 2 diabetic patients with advanced kidney disease will lead to preservation of kidney function.

DETAILED DESCRIPTION:
Diabetic kidney disease is the leading cause of new cases of kidney failure in the United States. In the kidneys of diabetic patients, there is accumulation of protein that leads to the formation of scar tissue and poor kidney function. Because of this many patients eventually require dialysis or kidney transplantation. A new investigational drug, pirfenidone, has been shown to be beneficial in a number of diseases in which scar formation leads to disease progression. It is our goal to examine whether pirfenidone is effective at stabilizing or reducing progressive diabetic kidney dysfunction.

ELIGIBILITY:
Inclusion

* Type 1 or type 2 diabetes
* Males and females greater than or equal to 18 years.
* Abnormal kidney function determined by glomerular filtration rate
* History of proteinuria
* Blood pressure controlled to <140/90 on anti-hypertensive medication

Exclusion

* Cancer, liver disease, hepatitis, HIV+
* History of heart attack, unstable angina, stroke or peptic ulcer in the past 6 months
* Pregnant or planning to become pregnant during the study period
* Other known kidney disease besides diabetic nephropathy
* Expect to begin dialysis or receive a kidney transplant within 1 year of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-06; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the change in renal function from baseline to the end of the study period (12 months). | 12 months

SECONDARY OUTCOMES:
% change in urine albumin excretion from baseline to end of study period. | 12 months
% change in levels of TGF-b1 in urine, plasma and serum from baseline to end of study period. | 12 months
• Determine the relationship between % change in TGF-b1 levels and the change in GFR | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Sharma, M.D., Principal Investigator — UCSD
Locations (3):
- United States (3):
  - National Institute of Diabetes and Digestive and Kidney Disease (NIDDK), Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - The Center for Diabetic Kidney Disease at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Sharma K, Ziyadeh FN, Alzahabi B, McGowan TA, Kapoor S, Kurnik BR, Kurnik PB, Weisberg LS. Increased renal production of transforming growth factor-beta1 in patients with type II diabetes. Diabetes. 1997 May;46(5):854-9. doi: 10.2337/diab.46.5.854. PMID 9133555
- [Background] Shimizu F, Fukagawa M, Yamauchi S, Taniyama M, Komemushi S, Margolin SB, Kurokawa K: Pirfenidone prevents the progression of irreversible glomerular sclerotic lesions in rats. Nephrology 3:315-322, 1997
- [Background] Shimizu T, Fukagawa M, Kuroda T, Hata S, Iwasaki Y, Nemoto M, Shirai K, Yamauchi S, Margolin SB, Shimizu F, Kurokawa K. Pirfenidone prevents collagen accumulation in the remnant kidney in rats with partial nephrectomy. Kidney Int Suppl. 1997 Dec;63:S239-43. PMID 9407470
- [Background] Iyer SN, Gurujeyalakshmi G, Giri SN. Effects of pirfenidone on transforming growth factor-beta gene expression at the transcriptional level in bleomycin hamster model of lung fibrosis. J Pharmacol Exp Ther. 1999 Oct;291(1):367-73. PMID 10490926
- [Background] McGowan T, Dunn SR, Sharma K: Treatment of db/db mice with pirfenidone leads to improved histology and serum creatinine. J Am Soc Nephrology 11:A2814, 2000
- [Background] Raghu G, Johnson WC, Lockhart D, Mageto Y. Treatment of idiopathic pulmonary fibrosis with a new antifibrotic agent, pirfenidone: results of a prospective, open-label Phase II study. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1061-9. doi: 10.1164/ajrccm.159.4.9805017. PMID 10194146